CLINICAL TRIAL: NCT01840969
Title: Association of Carotid Arterial Circumferential Strain With Left Ventricular Function and Hemodynamic Compromise During Off-pump Coronary Artery Bypass Surgery
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2011-0467
Record Dates: First submitted 2013-04-10; First posted 2013-04-26 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Three Vessel Coronary Artery Disease
Keywords: off-pump coronary artery bypass surgery; common carotid artery; speckle tracking analysis; peak strain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CAOD group: Single arm study group

SUMMARY:
This study is aimed to evaluate the association of common carotid artery circumferential strain with the echocardiographic parameters of left ventricular function and the degree of actual hemodynamic deterioration in patients undergoing multi-vessel off-pump coronary artery bypass with preserved left ventricular ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

1. three vessel coronary artery disease
2. sinus rhythm

Exclusion Criteria:

1. New York Heart Association functional class ≥3
2. known pulmonary hypertension
3. known valvular heart disease
4. serum creatinine ≥2.0 mg/dL
5. myocardial infarction within 1 week before the surgery
6. history of cerebral or peripheral arterial occlusive disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective multivessel off-pump coronary artery bypass surgery
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2011-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
TTE parameters | 1 day before the surgery
  TTE parameters: left ventricular ejection fraction, left atrial volume index, left ventricular mass, Sm, Em, E/Em

SECONDARY OUTCOMES:
change of intraoperative hemodynamic variables | from after induction of anesthesia, left circumflex artery grafting, and to sternum closure
  TTE parameters: left ventricular ejection fraction, left atrial volume index, left ventricular mass, Sm, Em, E/Em Carotid circumferential strain : Storage of transverse image of the right CCA at approximately 1cm proximal to the bifurcation, manual trace of luminal-intimal border and automatic tracking by frame-to-frame movement of ultrasound reflections (speckles) Hemodynamic variables: cardiac index and mixed venous oxygen saturation obtained from the pulmonary artery catheter and cardiac output monitoring devices

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University College of Medicine, Seoul, Seoul, South Korea